CLINICAL TRIAL: NCT03363633
Title: Randomized Trial of Perforator Vein Injection for Symptomatic Venous Disease
Brief Title: Perforator Vein Injection for Symptomatic Venous Disease
Acronym: Dillavou
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting
Sponsor: Ellen Dillavou (Other)
Collaborators: American College of Phlebology (Other)
Responsible Party: Sponsor-Investigator, Ellen Dillavou, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol #4
Record Dates: First submitted 2017-06-04; First posted 2017-12-06 (Actual); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Venous Disease
Keywords: Venous Ulceration; Refluxing Perforator Veins
MeSH Terms: conditions — Varicose Ulcer | interventions — Sodium Tetradecyl Sulfate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observation (No Intervention)
- Injection + Compression (Experimental)
  Interventions: Drug: sodium tetradecyl sulfate; Device: Compression
- Compression (Active Comparator)
  Interventions: Device: Compression

INTERVENTIONS:
Drug: sodium tetradecyl sulfate — Ultrasound-guided injection with sodium tetradecyl sulfate foam of refluxing perforating veins
  Arms: Injection + Compression
Device: Compression — 20-30 mmHg compression stockings
  Arms: Compression; Injection + Compression

SUMMARY:
The primary objective of this study is to compare two treatment strategies for symptomatic venous stasis disease with and without venous ulcer. These treatments are compression therapy alone vs. sclerotherapy of refluxing perforating veins with compression.

DETAILED DESCRIPTION:
Symptomatic venous disease is a widespread problem, affecting millions of patients per year, an estimated 1.0 - 1.5% of the population. This costs up to 1% of the total health care budget1-3. Venous problems account for almost 3000 patient visits in the UPP vascular surgery group per year. Although great progress has been made in venous stasis treatments there are still patients who suffer for many years with pain and ulceration due to venous disease. The investigators believe that venous hypertension is the underlying cause of venous ulceration. Three mechanisms leading to venous hypertension are well-recognized: superficial vein (great, accessory and small saphenous) incompetence; deep vein (common and superficial femoral, popliteal and tibial) reflux or obstruction; perforating vein incompetence. Patients with venous stasis and ulceration may have any or all of these conditions. Currently there are excellent treatments for superficial venous reflux, namely laser or radiofrequency ablation. Deep venous reflux therapy is still under investigation, with prosthetic valves in trial. However, compression is still the mainstay of therapy. The presence of deep venous reflux has been shown to have a significant effect on ulcer healing when perforator treatment has been investigated4. Refluxing perforator vein treatment is currently in flux, with the existing options of open surgery and subfascial endoscopic perforator surgery (SEPS) being the most tested options, but with significant wound complications and long hospital stays associated with both7. The investigators are proposing a prospective trial to evaluate percutaneous perforator thrombosis to achieve similar results with less morbidity.

The population targeted is patients with venous stasis or ulceration who either do not have demonstrable superficial reflux amenable to ablation, or have venous symptoms and ulceration despite treatment of incompetent superficial veins. When patients have refluxing perforating veins, there is debate on optimal treatment. Open and endoscopic ligation and compression therapy have all been tried with varying degrees of success and morbidity. The average rate of healing in venous ulcers is approximately .05 cm/wk 5,6, which has been shown to significantly improve after perforator ligation4, but with high morbidity. Ultrasound-guided injection of perforating veins is now performed, but with largely unknown benefits and consequences. The investigators propose a prospective, randomized trial of perforator injection with sodium tetradecyl sulfate (STS) foam vs. compression as a means of determining the efficacy and morbidity of perforator STS foam injection for symptomatic venous disease. The investigators currently utilize both methods of treatment in practice. Injections and compression or compression alone are chosen based on each patient's clinical scenario. STS is currently approved by the U.S. Food and Drug Administration for intravenous use.

ELIGIBILITY:
Inclusion Criteria:

* • The subject must be > 18 years of age, male or female

  * Subject must be willing and able to wear compression stockings
  * Subject must have refluxing perforating veins ≥ 3.0 mm in diameter at the calf level or distally in the affected leg.
  * Subject presents with ulceration or other symptoms of venous stasis including:

rash, swelling, pain, bleeding, recurrent cellulitis

• The subject must sign a written informed consent, prior to randomization, using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

* • Pregnancy

  * Known allergy to STS
  * Refusal to wear compression stocking
  * Untreated significant great or small saphenous reflux
  * Disseminated malignancy or other terminal condition where subject is expected to live less than 6 months.
  * Significant arterial disease (ABI < .8)
  * Buergers disease
  * Acute superficial thrombophlebitis
  * Phlebitis migrans
  * Acute cellulitis
  * Clinical evidence of active local or systemic infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen D Dillavou, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Shadyside Medical Building, Suite 307, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Cai PL, Hitchman LH, Mohamed AH, Smith GE, Chetter I, Carradice D. Endovenous ablation for venous leg ulcers. Cochrane Database Syst Rev. 2023 Jul 27;7(7):CD009494. doi: 10.1002/14651858.CD009494.pub3. PMID 37497816

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Responsible Party is no longer at University of Pittsburgh and has confirmed that the study data were lost. The only information available is the study was terminated for recruitment difficulty following enrollment of 12 participants overall, with no breakdown per study arm (source: final report submitted to the IRB).
Groups:
- All Arms: Participants were randomized to either compression stockings or perforator vein injection with sodium tetradecyl sulfate, plus compression stockings.
Period: Overall Study
Arm/Group | All Arms
Started | 12
Completed | 0 (See note in Pre-Assignment Details)
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: The Responsible Party is no longer at University of Pittsburgh and has confirmed that the study data were lost. The only information available is the study was terminated for recruitment difficulty following enrollment of 12 participants overall, with no breakdown per study arm (source: final report submitted to the IRB).
Arm/Group | All Arms
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] — Population: See note in Baseline Analysis Population Description
Sex: Female, Male [Count of Participants; unit: Participants] — Population: See note in Baseline Analysis Population Description

OUTCOME MEASURES:

1. Primary Outcome: Ulcer Healing
Description: Change in wound size, reported in square centimeters
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | All Arms
Number analyzed (Participants) | 0

2. Secondary Outcome: Venous Clinical Severity Score (VCSS)
Description: The VCSS includes nine criteria of chronic venous disease, each graded from 0 to 3 (0=absent, 1=mild, 2=moderate, 3=severe). Up to three points may be added for differences in background conservative therapy (compression and elevation). The scores are then added, with a maximum score of 30.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | All Arms
Number analyzed (Participants) | 0

3. Secondary Outcome: Injection Complications
Description: Number of participants experiencing venous thromboses from injections
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | All Arms
Number analyzed (Participants) | 0

4. Secondary Outcome: Compliance With Compression Therapy
Description: Number of participants who use compression therapy
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | All Arms
Number analyzed (Participants) | 0

5. Secondary Outcome: Ulcer Recurrence
Description: Number of participants with ulcers that reopen after initial closure
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | All Arms
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The Responsible Party is no longer at University of Pittsburgh and has confirmed that the study data were lost. The only information available is the study was terminated for recruitment difficulty following enrollment of 12 participants overall, with no breakdown per study arm (source: final report submitted to the IRB).
Arm/Group | All Arms
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No